CLINICAL TRIAL: NCT04338165
Title: Effect of Impact of PCSK9 Inhibitors on Coronary Microvascular Dysfunction in Patients With Atherosclerotic Cardiovascular Disease Proved by Myocardial Ischemia and Needing Coronarography : a Monocentric, Prospective, Randomized and Open-label Phase II Trial
Brief Title: Impact of PCSK9 Inhibitors on Coronary Microvascular Dysfunction in Patients With Atherosclerotic Cardiovascular Disease Proved by Myocardial Ischemia and Needing Coronarography
Acronym: MICROPROTECT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC19.186
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Proprotein convertase subtilisin/kexin type 9 inhibitor monoclonal antibody (Anti-PCSK9); Microvascular coronary dysfunction (CMVD); Coronary angioplasty; Cardiovascular imaging
MeSH Terms: conditions — Atherosclerosis | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evolocumab, 420 milligrams (Experimental): Single injection of 420 milligrams of evolocumab (REPATHA®) one month before coronary angiography and coronary microcirculation (IMR) measurement.
  Interventions: Drug: Evolocumab 140 MG/ML [Repatha]
- Control arm (No Intervention): Measurement of coronary microcirculation (IMR) during coronary angiography, without prior evolocumab injection.

INTERVENTIONS:
Drug: Evolocumab 140 MG/ML [Repatha] — 3 injections of evolocumab 140 milligrams performed within 30 minutes and self-administered (subcutaneously in the abdomen, thigh, or upper arm)
  Arms: Evolocumab, 420 milligrams

SUMMARY:
Proprotein convertase subtilisin/kexin type 9 inhibitor monoclonal antibodies (anti-PCSK9) significantly reduce the serum LDL-C level, leading to a regression of the coronary epicardial plaque demonstrated by intracoronary ultrasonography (IVUS), as well as cardiovascular events (CV) in patients with atherosclerotic CV disease treated with statin. The impact of PCSK9 inhibition on coronary microcirculation has never been assessed. However, microvascular coronary dysfunction (CMVD) is a powerful prognostic marker, irrespective of conventional CV risk factors, but also of the severity of the epicardial coronary involvement detected during coronary angiography. The investigators hypothesized that anti-PCSK9 would decrease CMVD, measured by the microcirculatory resistance index (MRI) during coronary angioplasty (Percutaneous coronary intervention, PCI) in patients with myocardial ischemia proved in myocardial scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, aged 40 to 85,
* More than 50 kilograms
* Defined at high cardiovascular risk according to European guidelines
* LDL-C level ≥ 0.7 g / L (biological assessment of less than 6 months)
* Having benefited from myocardial scintigraphy
* For which coronarography is indicated according to European guidelines
* Affiliated with social security,
* Signed informed consent form

Exclusion Criteria:

* Clinical presentation of unstable angina
* Patient whose state of physical or psychological health could compromise the obtaining of his informed consent and his compliance with the requirements of the protocol, with the study evaluation, procedures or completion.
* End stage disease (estimated survival of less than one year)
* Severe renal dysfunction, defined as an estimated creatinine clearance (MDRD) < 30 mL/min at screening
* Contra-indication to adenosin : hypersensitivity to active active substance or to any of the excipients, type II or III atrioventricular block or atrial disease (except for pacemaker users), long QT syndrome, severe arterial hypotension, acute heart failure, asthma and severe chronic obstructive pulmonary disease, unstable angina unstabilized by drug therapy, taking dipyridamole, aminophylline, theophylline or other xanthine base within 24 hours prior to adenosine administration
* Contra-indication to heparin: hypersensitivity to active substance or to any of the excipients, past heparin induced thrombopenia type II, haemorrhage.
* Prior Coronary Artery Bypass Graft Surgery (CABG)
* Prior myocardial infarction in the territory of ischemia
* New York Heart Association (NYHA) class III or IV, or last known left ventricular ejection fraction < 30%
* Known hemorrhagic stroke at any time
* Uncontrolled or recurrent ventricular tachycardia
* Uncontrolled hypertension defined as sitting systolic blood pressure (SBP) > 180 mmHg or diastolic BP (DBP) > 110 mmHg
* Actual use of PCSK9 inhibitor (evolocumab or others)
* Untreated or inadequately treated hyperthyroidism or hypothyroidism, controlled by biological assessment if needed, defined by thyroid stimulating hormone (TSH) < lower limit of normal (LLN) or > 1.5 times the upper limit of normal (ULN), respectively, and free thyroxine (T4) levels that are outside normal range at screening
* Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the ULN at screening
* Recipient of any major organ transplant (eg, lung, liver, heart, bone marrow, renal)
* Personal or family history of hereditary muscular disorders
* LDL apheresis within 12 months prior to randomization
* Creatinine Phosphokinase (CPK) > 5 ULN at screening
* Active infection or others active disease judge by investigator incompatible with the protocol completion
* Main known active infection including positive viral serology (Human Immunodeficiency Virus, Hepatitis B Virus and Hepatitis C Virus)
* Malignancy (except non-melanoma skin cancers, cervical in-situ carcinoma, breast ductal carcinoma in situ, or stage 1 prostate carcinoma) within the last 10 years
* Known sensitivity to evolocumab or their excipients to be administered during dosing or natural rubber / latex
* Patient likely to not be available to complete all protocol-required study visits or procedures.
* Patient in exclusion period of another study
* Woman able to procreate in the absence of highly effective contraception
* Persons referred to in Articles L1121-6 to L1121-8 of the French code of public health (this corresponds to all persons protected: pregnant or parturient women, breastfeeding mothers, persons deprived of liberty by judicial or administrative decision, persons subject to a legal protection measure).

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Impact of a PCSK9 inhibitor treatment on coronary microvascular dysfunction (CMVD) at 4 weeks in patients with atherosclerotic cardiovascular disease. | 4 weeks
  Index of microcirculatory resistance (IMR), measured during invasive coronary angiography and expressed in mmHg.s

SECONDARY OUTCOMES:
Impact of a PCSK9 inhibitor treatment on soluble VE-cadherin rate (sVE). | 4 weeks
  Measurement of sVE rate at baseline and four weeks after treatment with evolocumab or without treatment.
Impact of a PCSK9 inhibitor treatment on brachial hyperemia (HB). | 4 weeks
  Variation of the luminal diameter of the humeral artery with baseline and four weeks after treatment with evolocumab or without treatment.
Impact of a PCSK9 inhibitor treatment on the rate of peri-procedural myocardial infarction. | 4 weeks
  Troponin I level after PCI (peri-procedural myocardial pain will be defined as a post-angioplasty troponin level 10 times higher than the 99th percentile of troponin I).
Correlations between invasive and non-invasive (myocardial scintigraphy - myocardial perfusion entropy (MPE), concentration of sVE, HB) measurements of coronary microvascular dysfunction. | 4 weeks
  IMR, MPE, sVE and the variation of the luminal diameter of the humeral artery.
Correlations between the cardiovascular risk and the concentration of sVE and MPE. | 4 weeks
  Risk score, sVE rate and MPE.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Barone-Rochette, MD, PhD, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224
- [Background] Nicholls SJ, Puri R, Anderson T, Ballantyne CM, Cho L, Kastelein JJ, Koenig W, Somaratne R, Kassahun H, Yang J, Wasserman SM, Scott R, Ungi I, Podolec J, Ophuis AO, Cornel JH, Borgman M, Brennan DM, Nissen SE. Effect of Evolocumab on Progression of Coronary Disease in Statin-Treated Patients: The GLAGOV Randomized Clinical Trial. JAMA. 2016 Dec 13;316(22):2373-2384. doi: 10.1001/jama.2016.16951. PMID 27846344
- [Background] Clarkson P, Celermajer DS, Powe AJ, Donald AE, Henry RM, Deanfield JE. Endothelium-dependent dilatation is impaired in young healthy subjects with a family history of premature coronary disease. Circulation. 1997 Nov 18;96(10):3378-83. doi: 10.1161/01.cir.96.10.3378. PMID 9396430
- [Background] Suwaidi JA, Hamasaki S, Higano ST, Nishimura RA, Holmes DR Jr, Lerman A. Long-term follow-up of patients with mild coronary artery disease and endothelial dysfunction. Circulation. 2000 Mar 7;101(9):948-54. doi: 10.1161/01.cir.101.9.948. PMID 10704159
- [Background] Schachinger V, Britten MB, Zeiher AM. Prognostic impact of coronary vasodilator dysfunction on adverse long-term outcome of coronary heart disease. Circulation. 2000 Apr 25;101(16):1899-906. doi: 10.1161/01.cir.101.16.1899. PMID 10779454
- [Background] Halcox JP, Schenke WH, Zalos G, Mincemoyer R, Prasad A, Waclawiw MA, Nour KR, Quyyumi AA. Prognostic value of coronary vascular endothelial dysfunction. Circulation. 2002 Aug 6;106(6):653-8. doi: 10.1161/01.cir.0000025404.78001.d8. PMID 12163423
- [Background] Bugiardini R, Manfrini O, Pizzi C, Fontana F, Morgagni G. Endothelial function predicts future development of coronary artery disease: a study of women with chest pain and normal coronary angiograms. Circulation. 2004 Jun 1;109(21):2518-23. doi: 10.1161/01.CIR.0000128208.22378.E3. Epub 2004 May 10. PMID 15136498
- [Background] Taqueti VR, Hachamovitch R, Murthy VL, Naya M, Foster CR, Hainer J, Dorbala S, Blankstein R, Di Carli MF. Global coronary flow reserve is associated with adverse cardiovascular events independently of luminal angiographic severity and modifies the effect of early revascularization. Circulation. 2015 Jan 6;131(1):19-27. doi: 10.1161/CIRCULATIONAHA.114.011939. Epub 2014 Nov 16. PMID 25400060
- [Background] Fujii K, Kawasaki D, Oka K, Akahori H, Iwasaku T, Fukunaga M, Eguchi A, Sawada H, Masutani M, Lee-Kawabata M, Tsujino T, Ohyanagi M, Masuyama T. The impact of pravastatin pre-treatment on periprocedural microcirculatory damage in patients undergoing percutaneous coronary intervention. JACC Cardiovasc Interv. 2011 May;4(5):513-20. doi: 10.1016/j.jcin.2011.02.005. PMID 21596324
- [Background] Seidah NG, Awan Z, Chretien M, Mbikay M. PCSK9: a key modulator of cardiovascular health. Circ Res. 2014 Mar 14;114(6):1022-36. doi: 10.1161/CIRCRESAHA.114.301621. PMID 24625727
- [Background] Ding Z, Liu S, Wang X, Deng X, Fan Y, Sun C, Wang Y, Mehta JL. Hemodynamic shear stress via ROS modulates PCSK9 expression in human vascular endothelial and smooth muscle cells and along the mouse aorta. Antioxid Redox Signal. 2015 Mar 20;22(9):760-71. doi: 10.1089/ars.2014.6054. Epub 2015 Jan 8. PMID 25490141
- [Background] Ferri N, Tibolla G, Pirillo A, Cipollone F, Mezzetti A, Pacia S, Corsini A, Catapano AL. Proprotein convertase subtilisin kexin type 9 (PCSK9) secreted by cultured smooth muscle cells reduces macrophages LDLR levels. Atherosclerosis. 2012 Feb;220(2):381-6. doi: 10.1016/j.atherosclerosis.2011.11.026. Epub 2011 Nov 25. PMID 22176652
- [Background] Karagiannis AD, Liu M, Toth PP, Zhao S, Agrawal DK, Libby P, Chatzizisis YS. Pleiotropic Anti-atherosclerotic Effects of PCSK9 InhibitorsFrom Molecular Biology to Clinical Translation. Curr Atheroscler Rep. 2018 Mar 10;20(4):20. doi: 10.1007/s11883-018-0718-x. PMID 29525934
- [Background] Rochefort P, Chabaud S, Pierga JY, Tredan O, Brain E, Bidard FC, Schiffler C, Polena H, Khalil-Mgharbel A, Vilgrain I, Bachelot T. Soluble VE-cadherin in metastatic breast cancer: an independent prognostic factor for both progression-free survival and overall survival. Br J Cancer. 2017 Jan;116(3):356-361. doi: 10.1038/bjc.2016.427. Epub 2017 Jan 5. PMID 28056463
- [Background] Catapano AL, Graham I, De Backer G, Wiklund O, Chapman MJ, Drexel H, Hoes AW, Jennings CS, Landmesser U, Pedersen TR, Reiner Z, Riccardi G, Taskinen MR, Tokgozoglu L, Verschuren WMM, Vlachopoulos C, Wood DA, Zamorano JL, Cooney MT; ESC Scientific Document Group. 2016 ESC/EAS Guidelines for the Management of Dyslipidaemias. Eur Heart J. 2016 Oct 14;37(39):2999-3058. doi: 10.1093/eurheartj/ehw272. Epub 2016 Aug 27. No abstract available. PMID 27567407
- [Background] Ricchiuti V, Shear WS, Henry TD, Paulsen PR, Miller EA, Apple FS. Monitoring plasma cardiac troponin I for the detection of myocardial injury after percutaneous transluminal coronary angioplasty. Clin Chim Acta. 2000 Dec;302(1-2):161-70. doi: 10.1016/s0009-8981(00)00365-x. PMID 11074073
- [Background] Landmesser U, Chapman MJ, Stock JK, Amarenco P, Belch JJF, Boren J, Farnier M, Ference BA, Gielen S, Graham I, Grobbee DE, Hovingh GK, Luscher TF, Piepoli MF, Ray KK, Stroes ES, Wiklund O, Windecker S, Zamorano JL, Pinto F, Tokgozoglu L, Bax JJ, Catapano AL. 2017 Update of ESC/EAS Task Force on practical clinical guidance for proprotein convertase subtilisin/kexin type 9 inhibition in patients with atherosclerotic cardiovascular disease or in familial hypercholesterolaemia. Eur Heart J. 2018 Apr 7;39(14):1131-1143. doi: 10.1093/eurheartj/ehx549. No abstract available. PMID 29045644
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Fearon WF, Balsam LB, Farouque HM, Caffarelli AD, Robbins RC, Fitzgerald PJ, Yock PG, Yeung AC. Novel index for invasively assessing the coronary microcirculation. Circulation. 2003 Jul 1;107(25):3129-32. doi: 10.1161/01.CIR.0000080700.98607.D1. Epub 2003 Jun 23. PMID 12821539
- [Background] Yong AS, Layland J, Fearon WF, Ho M, Shah MG, Daniels D, Whitbourn R, Macisaac A, Kritharides L, Wilson A, Ng MK. Calculation of the index of microcirculatory resistance without coronary wedge pressure measurement in the presence of epicardial stenosis. JACC Cardiovasc Interv. 2013 Jan;6(1):53-8. doi: 10.1016/j.jcin.2012.08.019. PMID 23347861
- [Background] Ng MK, Yong AS, Ho M, Shah MG, Chawantanpipat C, O'Connell R, Keech A, Kritharides L, Fearon WF. The index of microcirculatory resistance predicts myocardial infarction related to percutaneous coronary intervention. Circ Cardiovasc Interv. 2012 Aug 1;5(4):515-22. doi: 10.1161/CIRCINTERVENTIONS.112.969048. Epub 2012 Aug 8. PMID 22874078